CLINICAL TRIAL: NCT02241421
Title: The Effect of the Knock Down of Gut Microbiota by Antibiotics on Parameters of Body Weight Control and Insulin Sensitivity
Brief Title: The Importance of the Gut Microbiota in Body Weight Control and Insulin Sensitivity
Acronym: ANTIBIOTICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 11-3-072
Record Dates: First submitted 2012-10-22; First posted 2014-09-16 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Obesity; Insulin Resistance
Keywords: Impaired glucose tolerance; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Hyperinsulinism; Lipid metabolism; Anti Bacterial Agents; Gastro Intestinal Tract
MeSH Terms: conditions — Obesity; Insulin Resistance; Glucose Intolerance; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Hyperinsulinism | interventions — Amoxicillin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): No intervention: Placebo 3x2 capsules per day during 7 consecutive days.
  Interventions: Other: Placebo
- Treatment Antibiotics: Amoxicillin (Experimental): Experimental: Amoxicillin (broad spectrum antibiotics) 1500 mg/day (3x2 capsules of 250 mg) during 7 consecutive days.
  Interventions: Drug: Amoxicillin
- Treatment Antibiotics: Vancomycin (Experimental): Experimental: Vancomycin (small spectrum antibiotics) 1500mg/day (3x2 capsules of 250 mg) during 7 consecutive days
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Amoxicillin
  Arms: Treatment Antibiotics: Amoxicillin
Drug: Vancomycin
  Other Names: Vancocin CP 250
  Arms: Treatment Antibiotics: Vancomycin
Other: Placebo
  Arms: Placebo

SUMMARY:
BACKGROUND: The relation between gut microbiota and obesity originates from animal studies, showing that the change of gut microbiota can induce changes in both insulin resistance and body composition. In addition, these studies have shown changes in gut permeability inducing a pro-inflammatory state, changes in adipose tissue function and inflammation, effects on energy harvesting and metabolism, skeletal muscle fatty acid partitioning and fat oxidation. Human data is lacking, although several studies suggested that the composition of the gut microbiota differs between lean and obese, and between diabetic and non-diabetic individuals.

OBJECTIVE: To provide insight in the physiological significance and underlying mechanisms involved in the relation between gut microbiota, energy balance and insulin sensitivity in overweight men with impaired glucose homeostasis.

DETAILED DESCRIPTION:
The view on the putative significance of gut microbiota in metabolism emerged from animal studies. Bäcked et al. showed that germ free mice had 40% less body fat compared to conventionally raised mice. Transplantation of a cecum-derived microbial community of conventional mice into germ free mice, resulted in a significant increase of body weight and insulin resistance within 2 weeks. Application of metagenomic techniques in leptin-deficient ob/ob mice showed a different proportion of bacteria belonging when compared to lean, wild-type or heterozygous mice, with a greater representation of Firmicutes and fewer Bacteroidetes. This obese gut microbiome showed an enrichment in genes involved in energy extraction from food, less energy left over in the faeces and higher contents of the short-chain fatty acids (SCFAs) propionate, acetate and butyrate in the cecum.

Furthermore, microbiota composition may alter gut permeability, and may play a role in the development of metabolic endotoxemia (inflammation) and related impairments in glucose metabolism. In addition, the gut microbiota may determine AMP-activated protein kinase (AMPK) levels in muscle and liver, thereby affecting fatty acid oxidation (substrate metabolism) and fat storage. However, underlying mechanisms are not completely understood.

Therefore, researchers within the Top Institute Food and Nutrition (TIFN) have designed a multidisciplinary project ('Microbiota, energy balance and metabolism'), to fill the unmet gap between gut microbiota and human energy metabolism. The current protocol is designed to clarify the role of the gut microbiota in host energy metabolism and insulin sensitivity, with the main focus on underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* male
* 35-70 years
* caucasian
* overweight/obese (BMI 25-35 kg/m2)
* insulin resistant (Homeostasis Model of Assessment - Insulin Resistance (HOMA_IR) > 2.2)
* impaired glucose tolerance (IGT: 2h plasma glucose during 75g Oral Glucose Tolerance Test(OGTT) 7.8-11.1 mmol/l) and/or impaired fasting glucose (plasma glucose ≥ 5.6 mmol/l)
* body weight stable for at least three months (±3 kg)

Exclusion Criteria:

* known allergic reaction to vancomycin, teicoplanin, amoxicillin and other β-lactam antibiotics (penicillins and cefalosporins) or related antibiotics
* diabetes mellitus
* hearing disorders
* cardiovascular disease
* kidney disease
* gastrointestinal disease
* cancer
* asthma or bronchitis
* liver malfunction
* major illness with a life expectancy < 5 years
* diseases affecting glucose tolerance (e.g. pheochromocytoma, Cushing's syndrome, acromegaly), - - use of antibiotics in the past 3 months
* plans to lose weight and participation in organized sports activities for >3 hours per week
* The use of β-blockers, lipid lowering-drugs, glucose-lowering agents (including all sulfonylureas, biguanides, α-glucosidase inhibitors, thiazolidinediones, repaglinide, nateglinide and insulin), anti-oxidants or chronic corticosteroids treatment (> 7 consecutive days of treatment)

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | up to two weeks
  Before and after the intervention, insulin sensitivity will be measured by using the hyperinsulinemic-euglycemic clamp technique including a glucose tracer to accurately quantify glucose fluxes at the whole body level. Glucose and Insulin levels will be determined.

SECONDARY OUTCOMES:
Fatty Acid Handling in the muscle | up to two weeks
  Because skeletal muscle is responsible for almost 80% of insulin-stimulated glucose disposal, and comprises up to 40% of total body mass, it can be considered to be a major tissue in the etiology of insulin resistance. Therefore, it is important to study the role of skeletal muscle substrate metabolism (fatty acid handling)in the context of this study. Fatty acids, glycerol, triacylglycerol and labelled palmitate in the chylomicron fraction will be measured.
Markers of inflammation | up to two weeks
  Low-grade inflammation seems to contribute to insulin resistance in obese insulin resistant subjects. Therefore, muscle and adipose tissue expression/secretion of inflammatory molecules (i.e. TNFα, IL-6) will be measured.
Energy expenditure | up to two weeks
  Indirect calorimetry measurements will be done to determine energy expenditure (O2 and CO2). While the gut microbiota plays an important role in nutrient metabolism and energy extraction from the diet, the determination of energy expenditure and energy content in faeces will provide important insight into the role of the gut microbiota in body weight regulation.
Microbiota composition and energy content in faecal samples | up to two weeks
  The composition of bacteria in the gut will be determined before and after intervention to link the composition to the primary and other secondary parameters. The energy content in the faeces will provide insight in the energy extraction capacity of the bacteria present.
Gut wall permeability | up to two weeks
  A proposed hypothesis is that gut permeability plays an important role in the induction of inflammation in obese insulin resistant subjects. A multi-sugar whole gut permeability assay will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen E Blaak, Prof.Dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] Reijnders D, Goossens GH, Hermes GDA, Smidt H, Zoetendal EG, Blaak EE. Short-Term Microbiota Manipulation and Forearm Substrate Metabolism in Obese Men: A Randomized, Double-Blind, Placebo-Controlled Trial. Obes Facts. 2018;11(4):318-326. doi: 10.1159/000492114. Epub 2018 Aug 9. PMID 30089301
- [Derived] Jocken JWE, Reijnders D, Canfora EE, Boekschoten MV, Plat J, Goossens GH, Blaak EE. Effects of gut microbiota manipulation on ex vivo lipolysis in human abdominal subcutaneous adipocytes. Adipocyte. 2018;7(2):106-112. doi: 10.1080/21623945.2018.1464366. Epub 2018 Apr 25. PMID 29693476